CLINICAL TRIAL: NCT06094335
Title: Influence of Virtual Reality Rehabilitation Training on Posture Control in Children With Autism Spectrum Disorders
Brief Title: Effect of Virtual Reality on Balance in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Professor of physical therapy, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRR
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Autism
Keywords: autism spectrum disorder; Biodex; Postural Control; Virtual Reality
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Study and control groups
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): Virtual reality plus traditional physical therapy
  Interventions: Device: Virtual reality rehabilitation; Other: Traditional physical therapy
- Control (Active Comparator): Traditional physical therapy
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Device: Virtual reality rehabilitation — Children in this group received Virtual Reality Rehabilitation plus traditional physical therapy
  Arms: Study
Other: Traditional physical therapy — Flexibility exercises, strengthening exercises, endurance exercises, and postural stability exercises

SUMMARY:
Children with ASD have poorer postural balance when compared to normal individuals. So, The aim of this study is to assess the effect of Virtual Reality on postural control in Autistic children

DETAILED DESCRIPTION:
Autism spectrum disorders are a collection of persistent neurodevelopmental disorders characterized by difficulties in social interactions, communication, and repetitive, stereotyped, and restricting behaviors. Movement problems can occur throughout infancy and are one of the early indications of autism. Furthermore, movement impairments are the most often observed nonverbal deficits in autistic children.

Postural stability is described as the capacity to maintain an upright posture by keeping the body's center of gravity over its base of support with little swaying or maximal steadiness, and it is considered a fundamental skill required for normal motor development.

Virtual Reality has been used in the field of balance rehabilitation and training because of its relatively low cost and enjoyment. Therefore, the purpose of this study was to study the effect of VR on balance in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Mild ASD

Exclusion Criteria:

* Taking medication affect motor
* Had a head injury, genetic disorder, blindness, fracture

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Static Balance | 12 weeks
  Change of overall postural sway scores using Biodex balance system
Functional Balance | 12 weeks
  Change in balance scores was measured using a pediatric balance scale. PBS collect scores for the 14 tasks assessed. The tasks are scored on a five-point scale (0, 1, 2, 3, or 4), with zero denoting an inability to perform the activity without assistance and four denoting the ability to perform the task with complete independence. Scores range from 0 to 56, with higher scores indicating better postural control

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdel Ghafar, Ph.D., Principal Investigator — Batterjee Medical College
Locations (1):
- Local Autism Center, Jeddah, Saudi Arabia